CLINICAL TRIAL: NCT00765726
Title: A Postauthorization Safety Surveillance Study Of Xyntha In Usual Care Settings
Brief Title: Study Evaluating The Safety Of Xyntha In Usual Care Settings
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: See termination reason in detailed description.
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 3082B2-4418; B1831003
Record Dates: First submitted 2008-10-02; First posted 2008-10-03 (Estimated); Results first posted 2012-01-20 (Estimated); Last update posted 2012-01-20 (Estimated); Status verified 2011-12

CONDITIONS: Hemophilia A
Keywords: hemophilia; hemophilia A; ReFacto; Xyntha; moroctocog alfa; bleeding disorder
MeSH Terms: conditions — Hemophilia A; Hemostatic Disorders | interventions — F8 protein, human; Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Moroctocog alfa(AF-CC) (Other)
  Interventions: Biological: Moroctocog alfa(AF-CC); Procedure: Blood draw for laboratory testing

INTERVENTIONS:
Biological: Moroctocog alfa(AF-CC) — Dosing is at the discretion of the investigator during the study
  Other Names: Xyntha
Procedure: Blood draw for laboratory testing — Hematology and Chemistry panels, Factor VIII inhibitor and recovery studies

SUMMARY:
The purpose of this study is to collect safety information associated with the use of Xyntha in a usual care setting. Upon meeting eligibility criteria, patients will be required to have approximately 5 study visits over a 2 year period. Procedures completed throughout the study include collection of vital signs, physical exams, and laboratory assessments. Patients will be required to complete an infusion log for each Xyntha infusion.

DETAILED DESCRIPTION:
The study was terminated on May 12, 2011 due to poor enrollment prospects and the study's similarity to another ongoing trial with ReFacto AF.

The termination of this study has no impact on subject safety or well being. The decision to terminate the trial was not based on any safety concerns.

ELIGIBILITY:
Inclusion Criteria:

* Male patients 12 years of age and older.
* Patients transitioned to Xyntha from other recombinant or plasma-derived FVIII replacement products.
* Treatment history of 150 or greater exposure days to any FVIII products prior to Enrollment visit.
* Negative inhibitor at screening or documentation of negative inhibitor titer within 6 weeks or less prior to study entry except for patients entering the study on immune tolerance induction therapy.

Exclusion Criteria:

* Bleeding disorder other than hemophilia A.
* Inhibitor titer greater than or equal to 0.6 BU during screening except for patients on immune tolerance induction therapy.
* Immunomodulatory therapy during screening period.
* Known hypersensitivity to hamster protein.

Min Age: 12 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2009-02; Primary Completion 2011-07 (Actual); Study Completion 2011-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (6):
- United States (5):
  - Pfizer Investigational Site, Los Angeles, California
  - Pfizer Investigational Site, Washington D.C., District of Columbia
  - Pfizer Investigational Site, Detroit, Michigan
  - Pfizer Investigational Site, East Lansing, Michigan
  - Pfizer Investigational Site, Dayton, Ohio
- Pfizer Investigational Site, Christchurch, New Zealand, New Zealand

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=3082B2-4418&StudyName=Study%20Evaluating%20The%20Safety%20Of%20Xyntha%20In%20Usual%20Care%20Settings

RESULTS

PARTICIPANT FLOW:
Groups:
- Xyntha: Xyntha [moroctocog alfa albumin free cell culture (AF-CC)] administered intravenously (IV) at a dose and frequency prescribed by the treating physician as per local standard of care for up to 2 years.
Period: Overall Study
Arm/Group | Xyntha
Started | 12
Completed | 3
Not Completed | 9
Not completed — Withdrawal by Subject | 1
Not completed — Discontinuation of study by sponsor | 8

BASELINE CHARACTERISTICS:
Arm/Group | Xyntha
Number analyzed (Participants) | 12
Age Continuous [Mean (Standard Deviation); unit: Years] | 30 (13.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 12

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Factor VIII (FVIII) Inhibitor Development
Description: FVIII inhibitor development was defined as an inhibitor titer of more than or equal to 0.6 Bethesda Units (BU) using the Nijmegen modification of the Bethesda assay and confirmed by the central laboratory.
Time Frame: Month 24 or early withdrawal
Population: Safety analysis population included all enrolled participants who had taken at least 1 dose of the study medication.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Xyntha
Number analyzed (Participants) | 12
Percentage of participants | 0.00 [0.00 to 0.27]

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | Xyntha
Serious Adverse Events (participants affected / at risk) | 2/12
Other Adverse Events (participants affected / at risk) | 9/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Xyntha (N=12)
Tooth impacted (Gastrointestinal disorders) | 1
Therapeutic response decreased (General disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Xyntha (N=12)
Nausea (Gastrointestinal disorders) | 3
Vomiting (Gastrointestinal disorders) | 2
Constipation (Gastrointestinal disorders) | 1
Dental caries (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 1
Tongue discolouration (Gastrointestinal disorders) | 1
Toothache (Gastrointestinal disorders) | 1
Corneal abrasion (Injury, poisoning and procedural complications) | 1
Head injury (Injury, poisoning and procedural complications) | 1
Incision site hypoaesthesia (Injury, poisoning and procedural complications) | 1
Procedural pain (Injury, poisoning and procedural complications) | 1
Stress fracture (Injury, poisoning and procedural complications) | 1
Tooth fracture (Injury, poisoning and procedural complications) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 3
Arthropathy (Musculoskeletal and connective tissue disorders) | 1
Osteomalacia (Musculoskeletal and connective tissue disorders) | 1
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 1
Joint swelling (Musculoskeletal and connective tissue disorders) | 1
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1
Pain in jaw (Musculoskeletal and connective tissue disorders) | 1
Ear infection (Infections and infestations) | 1
Herpes zoster (Infections and infestations) | 1
Influenza (Infections and infestations) | 1
Sinusitis (Infections and infestations) | 1
Upper respiratory tract infection (Infections and infestations) | 1
Infusion site phlebitis (General disorders) | 1
Non-cardiac chest pain (General disorders) | 1
Haematuria (Renal and urinary disorders) | 1
Urinary retention (Renal and urinary disorders) | 1
Blister (Skin and subcutaneous tissue disorders) | 1
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1
Gynaecomastia (Reproductive system and breast disorders) | 1
Painful erection (Reproductive system and breast disorders) | 1
Palpitations (Cardiac disorders) | 1
Fanconi syndrome (Congenital, familial and genetic disorders) | 1
Ear pain (Ear and labyrinth disorders) | 1
Biliary dilatation (Hepatobiliary disorders) | 1
Body temperature increased (Investigations) | 1
Varicose vein (Vascular disorders) | 1
Procedural site reaction (Injury, poisoning and procedural complications) | 1

LIMITATIONS AND CAVEATS:
The study was discontinued because the sponsor had ongoing studies collecting similar safety data.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.